CLINICAL TRIAL: NCT00020631
Title: A Pilot Study Of Pirfenidone For The Treatment Of Radiation-Induced Fibrosis
Brief Title: Pirfenidone in Treating Patients With Fibrosis Caused by Radiation Therapy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000068675; NCI-01-C-0143; NCT00014924 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-04

CONDITIONS: Radiation Fibrosis
Keywords: radiation fibrosis
MeSH Terms: conditions — Radiation Fibrosis Syndrome | interventions — pirfenidone

INTERVENTIONS:
Drug: pirfenidone

SUMMARY:
RATIONALE: Pirfenidone may prevent or lessen fibrosis caused by radiation therapy.

PURPOSE: Pilot trial to study the effectiveness of pirfenidone in preventing or lessening fibrosis in patients who have undergone radiation therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and therapeutic efficacy of pirfenidone in cancer patients with radiation-induced fibrosis.

OUTLINE: Patients receive oral pirfenidone 3 times daily. Treatment continues for up to 2 years in the absence of disease progression or unacceptable toxicity.

Principal functional abilities are assessed at baseline, every 3 months, and at termination of therapy.

PROJECTED ACCRUAL: A total of 10-25 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Regional post-radiation fibrosis of a specific body area (e.g., neck, back, or extremities)

  * At least moderate impairment in at least 1 of the following principal functional abilities:

    * Range of motion
    * Strength
    * Edema
    * Swallowing
* Prior radiation for cancer received more than 6 months ago
* No evidence of recurrent or metastatic cancer
* No history of collagen vascular disease
* No positive antinuclear antibody

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Hepatitis B and C negative

Renal:

* Not specified

Other:

* HIV negative
* No evidence of second primary cancer
* No life-threatening situation requiring rehabilitation intervention
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent anticancer immunotherapy

Chemotherapy:

* No concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* See Disease Characteristics
* No concurrent anticancer radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent anticancer investigational agents
* Stable doses of medicine (e.g., non-steroidal anti-inflammatory drugs) currently being taken are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Camphausen, MD, Principal Investigator — NCI - Radiation Oncology Branch; ROB
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States